CLINICAL TRIAL: NCT06541561
Title: Efficacy of Transcutaneous Electrical Acupoint Stimulation on Postoperative Pain and Recovery in Patients Undergoing Pancreatectomy: a Prospective, Randomized Controlled Trial
Brief Title: Efficacy of TEAS on Postoperative Pain and Recovery in Patients Undergoing Pancreatectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024HX0803
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients who meet the enrollment criteria will be randomized 1:1 to either the transcutaneous electrical acupoint stimulation (TEAS) or the sham groups using a computer-generated random number table. After the randomization, use the opaque envelope, hide each group envelope into an opaque envelope, the envelope outside the code, will be sealed to the researcher, when the study, if the inclusion criteria, then open the corresponding numbered envelope, and intervene according to the group scheme in the envelope.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding of participants will be maintained throughout the observation period. The sham group will receive electrode attachment but without stimulation, Throughout the study, for adequate blinding, an opaque tape will be applied to the patient's skin above the electrodes, and the patient's target acupoints will be wrapped in a blanket. All patients will be informed that they might or might not feel a tingling sensation around the acupoints when the TEAS device is working. The patients should not be unblinded until the statistical analysis of the study data is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TEAS group (Experimental): In the TEAS group, the acupoints are bilateral neiguan (PC6), Zusanli (ST 36), Hegu (L14) and Waiguan (SJ5) acupoints. The treatment will consist of two phases: a 30-minute stimulation administered 30 minutes before anesthesia induction, and a 30-minute stimulation session once daily on postoperative days 1, 2, and 3. The stimulation intensity will be adjusted in accordance with the maximal level tolerated by each patient. Patients in the sham group will receive electrode attachment but without stimulation.
  Interventions: Device: transcutaneous electrical acupoint stimulation
- sham group (Sham Comparator): Patients in the sham group will receive electrode attachment but without stimulation.
  Interventions: Device: sham transcutaneous electrical acupoint stimulation

INTERVENTIONS:
Device: transcutaneous electrical acupoint stimulation — Patients in the TEAS group, the acupoints are bilateral neiguan (PC6), Zusanli (ST 36), Hegu (L14) and Waiguan (SJ5) acupoints. The treatment will consist of two phases: a 30-minute stimulation administered 30 minutes before anesthesia induction, and a 30-minute stimulation session once daily on postoperative days 1, 2, and 3. The stimulation intensity will be adjusted in accordance with the maximal level tolerated by each patient. Patients in the sham group will receive electrode attachment but without stimulation.
  Arms: TEAS group
Device: sham transcutaneous electrical acupoint stimulation — Patients in the sham group will receive electrode attachment but without stimulation.
  Arms: sham group

SUMMARY:
The purpose of this study is to access the effect of transcutaneous electrical acupoint stimulation on postoperative pain in patients undergoing pancreatectomy

DETAILED DESCRIPTION:
Patients who meet the enrollment criteria will be randomized 1:1 to either the transcutaneous electrical acupoint stimulation (TEAS) or the sham groups. In the TEAS group, the acupoints are bilateral neiguan (PC6), Zusanli (ST 36), Hegu (L14) and Waiguan (SJ5) acupoints. The treatment will consist of two phases: a 30-minute stimulation administered 30 minutes before anesthesia induction, and a 30-minute stimulation session once daily on postoperative days 1, 2, and 3. The stimulation intensity will be adjusted in accordance with the maximal level tolerated by each patient. Patients in the sham group will receive electrode attachment but without stimulation.

ELIGIBILITY:
Inclusion Criteria:

Age 18-80 years old; ASA physical status class I - III; Patients scheduled for pancreatectomy.

Exclusion Criteria:

Have a history of epilepsy; Rash or local infection over the acupoint stimulation skin area; Pregnancy or breastfeeding; Mental retardation, psychiatric, or neurological disease; Inability to comprehend the numeric rating scale (NRS); Implantation of a cardiac pacemaker, cardioverter, or defibrillator; Chronic opioid use; Metastases in other organs; Have a history of Transcutaneous Electrical Acupuncture Stimulation (TEAS) or electroacupuncture treatment in the past or recently；

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-07-16 (Estimated); Primary Completion 2026-09-02 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
highest NRS pain score for movement-evoked pain (defined as deep breathing or forced coughing three times) during 72 hours postoperatively. | Up to 72 hours postoperatively
  The pain is evaluated using numerical rating scale(NRS). NRS scores range from 0 to 10 points, with 0 points representing no pain, and 10 points representing the strongest pain.

SECONDARY OUTCOMES:
the highest NRS pain score at rest during 72 h postoperatively | Up to 72 hours postoperatively
  The pain is evaluated using numerical rating scale(NRS). NRS scores range from 0 to 10 points, with 0 points representing no pain, and 10 points representing the strongest pain.
The cumulative morphine consumption at 24, 48, and 72 hours postoperatively. | Up to 72 hours postoperatively
  Postoperative opioid use is reported as morphine milligram equivalents, calculated using the Practical Pain Management calculator
The incidence of postoperative nausea and vomiting during the first 24,48,72 hours. | Up to 72 hours postoperatively
  We considered it PONV if patients felt any nausea or had any vomiting.
The incidence of a composite of postoperative pulmonary complications during hospitalization. | Up to 7 days postoperatively
  Defined as positive if any component developed before discharge after surgery; These complications included respiratory infection, respiratory failure, pleural effusion, atelectasis, pneumothorax, bronchospasm, or aspiration pneumonitis loading dose, during hospitalization after surgery.
Quality of Recovery Scale Score at 24, 48, and 72 hours after surgery. | Up to 3 days postoperatively
  The global QoR-15 score ranges from 0 to 150 and is categorized as five quality of recovery dimensions, including physical comfort (5 items), emotional state (4 items), psychological support (2 items), physical independence (2 items), and pain (2 items). Each piece is graded using an 11-point Likert scale. The QoR is classified according to the QoR-15 score as excellent (QoR-15 > 135), good (122 ≤ QoR-15 ≤ 135), moderate (90 ≤ QoR-15 ≤ 121) and poor (QoR-15 < 90).
The postoperative sleep quality score | Up to 3 days postoperatively
  Postoperative sleep quality was evaluated using the Athens Insomnia Scale (AIS). The AIS consists of 8 items: waking up at night, sleep induction, final awakening, total sleep duration, sleep quality, well-being, functional ability, and daytime sleepiness. The AIS score ranges from 0 to 24 points, and a total score of 6 points or higher indicates a diagnosis of insomnia
The plasma levels of C-reactive protein (CRP), procalcitonin (PCT), beta-endorphin, serotonin (5-HT), interleukin-2 (IL-2), interleukin-6 (IL-6), and tumor necrosis factor-alpha (TNF-α) on the 1st, 3rd, and 5th postoperative days | Up to 5 days postoperatively]
  Peripheral blood C-reactive protein (CRP), procalcitonin (PCT), beta-endorphin, serotonin (5-HT), interleukin-2 (IL-2), interleukin-6 (IL-6), and tumor necrosis factor-alpha (TNF-α) are measured at the 1st, 3rd, and 5th postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Luo Fengming, PhD, Principal Investigator — West China Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu J, Chen J, Tang Q, Zhou L. Efficacy of perioperative transcutaneous electrical acupoint stimulation on postoperative pain and recovery in patients undergoing pancreatectomy: a study protocol for a randomized controlled trial. Trials. 2025 Dec 31. doi: 10.1186/s13063-025-09386-5. Online ahead of print. PMID 41469720